CLINICAL TRIAL: NCT01797978
Title: Infusion of Methylene Blue in Severe Sepsis and Septic Shock: Randomized, Single Blinded
Brief Title: Methylene Blue in Severe Sepsis and Septic Shock
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1210/173-002
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Sepsis; Septic shock; Methylene blue
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous methylene blue administration (Experimental): 2mg/kg IV bolus followed by 0.5mg/kg/hr slow infusion for 6hrs
  Interventions: Drug: Intravenous methylene blue administration
- Placebo (Placebo Comparator): Normal saline administration instead of methylene blue
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous methylene blue administration — Initial history taking and physical examination --> enrollment --> 2mg/kg IV bolus followed by 0.5mg/kg/hr slow infusion of methylene blue for 6hrs
  Other Names: methylene blue administration; MB administration
  Arms: Intravenous methylene blue administration
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is to see whether the intravenous administration of methylene blue improves the outcome in severe sepsis and septic shock.

DETAILED DESCRIPTION:
The mortality of septic shock is still high ranging from 30 to 50%. Vasopressor is the main part in managing septic shock, but the choice of vasopressor is still under-investigated, and area of uncertainty.

The response to vasopressor is sometimes unsatisfactory, and in that case, the outcome of the patients is poor.

Recently, small size clinical trial has investigated the effect of methylene blue (MB), and showed promising results. However, large sized phase III trial has not been performed yet.

Large sized phase III clinical trial is needed to establish the effect of MB in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock meeting the criteria of 2012 surviving sepsis campaign
* Need the norepinephrine of over 0.2microgram/kg/min

Exclusion Criteria:

* Pregnancy
* Less than 18 years old
* Terminal cancer patients
* Declined consents
* glucose-6-phosphate dehydrogenase deficiency
* Medication of Serotonin modulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | within 28 days of diagnosis

SECONDARY OUTCOMES:
Vasopressor dependent period | within 28 days of diagnosis
Vasopressor index | with in 28 days of diagnosis
Change of cardiac output (CO) and systemic vascular resistance (SVR) | with in 28 days of diagnosis
  EV1000 (Edwards inc.) will be used to see the cardiac output and systemic vascular resistance.
Length of stay in ICU (LOSICU) | with in 28 days of diagnosis
LOS in hospital | with in 28 days of diagnosis
In hospital mortality | with in 28 days of diagnosis
Multiple organ failure (SOFA) | with in 28 days of diagnosis
NO level | before and after infusion of MB, 24hrs, 48hrs later
Cytokine level (IL-6, 10, tumor necrosis factor -alpha) | before and after infusion of MB, 24hrs, 48hrs later

CONTACTS AND LOCATIONS:
Overall Officials: Kyuseok Kim, MD, Study Director — Professor, department of emergency medicine
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Kyeongi-do
  - Seoul National University Hospital, Seoul
  - SMG - SNU Boramae Medical Center, Seoul